CLINICAL TRIAL: NCT03297034
Title: Swiss Childhood Cancer Survivor Study (SCCSS)
Brief Title: Swiss Childhood Cancer Survivor Study
Acronym: SCCSS
Status: Recruiting | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: Swiss Pediatric Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: SCCSS
Record Dates: First submitted 2017-09-20; First posted 2017-09-29 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Childhood Cancer
Keywords: Late effects; Childhood cancer survivors; Swiss Childhood Cancer Registry; Europe
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The SCCSS is designed to investigate which long-term effects childhood cancer and its treatment have on survivors, and includes those who were under 20 years when they were diagnosed. The SCCSS explores childhood cancer survivors' quality of life, the health care received by childhood cancer survivors during follow-up care, the effects of medication, somatic and psychosocial health issues, how childhood cancer survivors take care of their own health including health behaviors, and also collects demographic details like family background, education and profession. To learn more about these topics, the investigators send questionnaires to childhood or adolescent cancer survivors. The investigators use the results to inform physicians and patients, and to improve treatment of childhood cancer and follow-up.

DETAILED DESCRIPTION:
The SCCSS is designed to investigate which long-term effects childhood cancer and its treatment have on survivors, and includes those who were under 20 years when they were diagnosed. The SCCSS explores childhood cancer survivors' quality of life, the health care received by childhood cancer survivors during follow-up care, the effects of medication, somatic and psychosocial health issues, how childhood cancer survivors take care of their own health including health behaviors, and also collects demographic details like family background, education and profession. To learn more about these topics, the investigators send questionnaires to childhood or adolescent cancer survivors. The investigators use the results to inform physicians and patients, and to improve treatment of childhood cancer and follow-up.

Background: Therapies have improved so much in the past decades that more than 80% of children and adolescents now survive cancer. This means that the population of long-term childhood cancer survivors is growing. Since cancer and its treatments may later have adverse effects, it is important to track and improve survivor health and quality of life. Comprehensive data on the burden of late effects of childhood cancer or risk factors for late effects was not available, and so Switzerland set up the SCCSS to increase knowledge and improve the quality of care and follow-up.

Objectives: The SCCSS investigates long-term outcomes of survivors of childhood and adolescent cancer, and the incidence and spectrum of various somatic and psychosocial outcomes including late mortality, second primary malignancies, somatic health and medication, mental health, educational achievements, health-related quality of life, and the association of these outcomes with risk factors like tumor, treatment modalities, and demographic characteristics. The SCCSS also investigates how health-care is provided, and how long-term childhood cancer survivors take care of their health inducing health behaviors.

Methods: All Swiss residents who were diagnosed with cancer at age <20 years, have survived at least 5 years since cancer diagnosis, received a detailed questionnaire. The investigators added data from general practitioners and hospital records. To compare survivors with the general population, they also send the questionnaire to the siblings of childhood cancer survivors. Since 2025 we ask participants of the SCCSS if they are interested in wearing an accelerometer for one week to track the amount of time they spend moving, sitting and sleeping (SCCSS-Activity).

Rationale and significance: The data collected by the SCCSS allows the investigators to study long-term outcomes of Swiss childhood cancer survivors. The SCCSS helps to learn more about the incidence of late effects and their risk factors. It also allows to summarize the current state of care in Switzerland. Since early diagnosis can prevent or mitigate many late effects, tracking them will help to improve the health of current and future childhood cancer survivors.

Current status of the SCCSS: From 2008-2025, the investigators have contacted 6487 childhood cancer survivors diagnosed between 1976-2019 and 2074 of their siblings. The investigators contact new 5-year childhood cancer survivors at regular intervals, and continuously analyse and publish data and findings. By 2022, the investigators have contacted 3443 childhood cancer survivors for a follow-up questionnaire and will continue with this at regular intervals.

Current status of the SCCSS-Activity: From 2025, the investigators have asked 319 participants of the SCCSS if they are interested in participating in the SCCSS-Activity.

Funding: Swiss Cancer League/ Swiss Cancer Research (Grant No: KLS/KFS-4825-01-2019), Stiftung für krebskranke Kinder (Regio basiliensis) and Kinderkrebshilfe Schweiz.

ELIGIBILITY:
Inclusion Criteria:

* Who were diagnosed with cancer at age <20 years
* Who have survived at least 5 years after cancer diagnosis
* Who were Swiss residents when they were diagnosed, and
* Who gave informed consent

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Childhood cancer survivors: All living individuals who were diagnosed with cancer at age <20 years, have survived at least 5 years after cancer diagnosis, and who were Swiss residents when they were diagnosed.
  Siblings: brothers and sisters of childhood cancer survivors.
Sampling Method: Non-Probability Sample
Enrollment: 4076 (Estimated)
Dates: Start 2007-01-01 (Actual); Primary Completion 2050-01 (Estimated); Study Completion 2050-01 (Estimated)

PRIMARY OUTCOMES:
Long-term outcomes of survivors of childhood and adolescent cancer | Baseline medical information and questionnaire data collection among those who survived at least 5 years, follow-up data collection at regular intervals (+/- every 5 years, 40 years) afterwards.
  Incidence and spectrum of various somatic and psychosocial outcomes including describing the cause-specific long-term mortality, the number of patients with second primary malignancies and somatic health effects, and describe medication use, mental health status, educational achievements, and health-related quality of life of childhood cancer survivors as assessed by questionnaires and data from the Swiss Childhood Cancer Registry.

SECONDARY OUTCOMES:
Risk factors of long-term outcomes of survivors of childhood and adolescent cancer | Baseline medical information and questionnaire data collection among those who survived at least 5 years, follow-up data collection at regular intervals (+/- every 5 years, 40 years) afterwards.
  Association of long-term outcomes with risk factors like tumour, treatment modalities, and demographic characteristics as assessed by questionnaires and data from the Swiss Childhood Cancer Registry.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia E Kuehni, Prof., Study Director — Institute of Social and Preventive Medicine (ISPM), Univeristy of Bern
Locations (1):
- Institute of Social and Preventive Medicine (ISPM), University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kasteler R, Weiss A, Schindler M, Sommer G, Latzin P, von der Weid NX, Ammann RA, Kuehni CE; Swiss Pediatric Oncology Group (SPOG). Long-term pulmonary disease among Swiss childhood cancer survivors. Pediatr Blood Cancer. 2018 Jan;65(1). doi: 10.1002/pbc.26749. Epub 2017 Sep 4. PMID 28868646
- [Result] Rueegg CS, Gianinazzi ME, Michel G, Zwahlen M, von der Weid NX, Kuehni CE; and the Swiss Paediatric Oncology Group (SPOG). No evidence of response bias in a population-based childhood cancer survivor questionnaire survey - Results from the Swiss Childhood Cancer Survivor Study. PLoS One. 2017 May 2;12(5):e0176442. doi: 10.1371/journal.pone.0176442. eCollection 2017. PMID 28463966
- [Result] Weiss A, Sommer G, Kuonen R, Scheinemann K, Grotzer M, Kompis M, Kuehni CE; Swiss Paediatric Oncology Group (SPOG). Validation of questionnaire-reported hearing with medical records: A report from the Swiss Childhood Cancer Survivor Study. PLoS One. 2017 Mar 23;12(3):e0174479. doi: 10.1371/journal.pone.0174479. eCollection 2017. PMID 28333999
- [Result] Belle F, Wengenroth L, Weiss A, Sommer G, Beck Popovic M, Ansari M, Bochud M, Kuehni C; Swiss Paediatric Oncology Group (SPOG). Low adherence to dietary recommendations in adult childhood cancer survivors. Clin Nutr. 2017 Oct;36(5):1266-1274. doi: 10.1016/j.clnu.2016.08.012. Epub 2016 Oct 20. PMID 28277304
- [Result] Weiss A, Sommer G, Kasteler R, Scheinemann K, Grotzer M, Kompis M, Kuehni CE; Swiss Pediatric Oncology Group (SPOG). Long-term auditory complications after childhood cancer: A report from the Swiss Childhood Cancer Survivor Study. Pediatr Blood Cancer. 2017 Feb;64(2):364-373. doi: 10.1002/pbc.26212. Epub 2016 Sep 21. PMID 27650356
- [Result] Wengenroth L, Sommer G, Schindler M, Spycher BD, von der Weid NX, Stutz-Grunder E, Michel G, Kuehni CE; Swiss Paediatric Oncology Group (SPOG). Income in Adult Survivors of Childhood Cancer. PLoS One. 2016 May 23;11(5):e0155546. doi: 10.1371/journal.pone.0155546. eCollection 2016. PMID 27213682
- [Result] Wengenroth L, Gianinazzi ME, Rueegg CS, Luer S, Bergstraesser E, Kuehni CE, Michel G. Health-related quality of life in young survivors of childhood cancer. Qual Life Res. 2015 Sep;24(9):2151-61. doi: 10.1007/s11136-015-0961-3. Epub 2015 Mar 18. PMID 25784561
- [Result] Wengenroth L, Rueegg CS, Michel G, Gianinazzi ME, Essig S, von der Weid NX, Grotzer M, Kuehni CE; Swiss Paediatric Oncology Group SPOG. Concentration, working speed and memory: cognitive problems in young childhood cancer survivors and their siblings. Pediatr Blood Cancer. 2015 May;62(5):875-82. doi: 10.1002/pbc.25396. Epub 2015 Feb 2. PMID 25645276
- [Result] Wengenroth L, Rueegg CS, Michel G, Essig S, Ammann RA, Bergstraesser E, Kuehni CE; Swiss Paediatric Oncology Group (SPOG). Life partnerships in childhood cancer survivors, their siblings, and the general population. Pediatr Blood Cancer. 2014 Mar;61(3):538-45. doi: 10.1002/pbc.24821. Epub 2013 Oct 18. PMID 24136901
- [Result] Gianinazzi ME, Rueegg CS, von der Weid NX, Niggli FK, Kuehni CE, Michel G; Swiss Paediatric Oncology Group (SPOG). Mental health-care utilization in survivors of childhood cancer and siblings: the Swiss childhood cancer survivor study. Support Care Cancer. 2014 Feb;22(2):339-49. doi: 10.1007/s00520-013-1976-3. Epub 2013 Oct 1. PMID 24081625
- [Result] Gianinazzi ME, Essig S, Rueegg CS, von der Weid NX, Brazzola P, Kuehni CE, Michel G; Swiss Paediatric Oncology Group (SPOG). Information provision and information needs in adult survivors of childhood cancer. Pediatr Blood Cancer. 2014 Feb;61(2):312-8. doi: 10.1002/pbc.24762. Epub 2013 Sep 9. PMID 24019260
- [Result] Rueegg CS, Gianinazzi ME, Rischewski J, Beck Popovic M, von der Weid NX, Michel G, Kuehni CE. Health-related quality of life in survivors of childhood cancer: the role of chronic health problems. J Cancer Surviv. 2013 Dec;7(4):511-22. doi: 10.1007/s11764-013-0288-4. Epub 2013 Jun 20. PMID 23784593
- [Result] Rueegg CS, Gianinazzi ME, Michel G, von der Weid NX, Bergstraesser E, Kuehni CE; Swiss Paediatric Oncology Group (SPOG). Do childhood cancer survivors with physical performance limitations reach healthy activity levels? Pediatr Blood Cancer. 2013 Oct;60(10):1714-20. doi: 10.1002/pbc.24595. Epub 2013 May 16. PMID 23681516
- [Result] Gianinazzi ME, Rueegg CS, Wengenroth L, Bergstraesser E, Rischewski J, Ammann RA, Kuehni CE, Michel G; for Swiss Pediatric Oncology Group (SPOG). Adolescent survivors of childhood cancer: are they vulnerable for psychological distress? Psychooncology. 2013 Sep;22(9):2051-8. doi: 10.1002/pon.3249. Epub 2013 Feb 11. PMID 23401292
- [Result] Rueegg CS, Michel G, Wengenroth L, von der Weid NX, Bergstraesser E, Kuehni CE; Swiss Paediatric Oncology Group (SPOG). Physical performance limitations in adolescent and adult survivors of childhood cancer and their siblings. PLoS One. 2012;7(10):e47944. doi: 10.1371/journal.pone.0047944. Epub 2012 Oct 17. PMID 23082232
- [Result] Kuehni CE, Rueegg CS, Michel G, Rebholz CE, Strippoli MP, Niggli FK, Egger M, von der Weid NX; Swiss Paediatric Oncology Group (SPOG). Cohort profile: the Swiss childhood cancer survivor study. Int J Epidemiol. 2012 Dec;41(6):1553-64. doi: 10.1093/ije/dyr142. Epub 2011 Oct 27. No abstract available. PMID 22736394
- [Result] Essig S, von der Weid NX, Strippoli MP, Rebholz CE, Michel G, Rueegg CS, Niggli FK, Kuehni CE; Swiss Pediatric Oncology Group (SPOG). Health-related quality of life in long-term survivors of relapsed childhood acute lymphoblastic leukemia. PLoS One. 2012;7(5):e38015. doi: 10.1371/journal.pone.0038015. Epub 2012 May 25. PMID 22662262
- [Result] Rueegg CS, von der Weid NX, Rebholz CE, Michel G, Zwahlen M, Grotzer M, Kuehni CE; Swiss Paediatric Oncology Group (SPOG). Daily physical activities and sports in adult survivors of childhood cancer and healthy controls: a population-based questionnaire survey. PLoS One. 2012;7(4):e34930. doi: 10.1371/journal.pone.0034930. Epub 2012 Apr 10. PMID 22506058
- [Result] Rebholz CE, Kuehni CE, Strippoli MP, Rueegg CS, Michel G, Hengartner H, Bergstraesser E, von der Weid NX; Swiss Pediatric Oncology Group (SPOG). Alcohol consumption and binge drinking in young adult childhood cancer survivors. Pediatr Blood Cancer. 2012 Feb;58(2):256-64. doi: 10.1002/pbc.23289. Epub 2011 Aug 29. PMID 22162398
- [Result] Kuehni CE, Strippoli MP, Rueegg CS, Rebholz CE, Bergstraesser E, Grotzer M, von der Weid NX, Michel G; Swiss Pediatric Oncology Group (SPOG). Educational achievement in Swiss childhood cancer survivors compared with the general population. Cancer. 2012 Mar 1;118(5):1439-49. doi: 10.1002/cncr.26418. Epub 2011 Aug 5. PMID 21823113
- [Result] Rebholz CE, von der Weid NX, Michel G, Niggli FK, Kuehni CE; Swiss Pediatric Oncology Group (SPOG). Follow-up care amongst long-term childhood cancer survivors: a report from the Swiss Childhood Cancer Survivor Study. Eur J Cancer. 2011 Jan;47(2):221-9. doi: 10.1016/j.ejca.2010.09.017. Epub 2010 Oct 11. PMID 20943372
- [Result] Michel G, Kuehni CE, Rebholz CE, Zimmermann K, Eiser C, Rueegg CS, von der Weid NX; Swiss Paediatric Oncology Group (SPOG). Can health beliefs help in explaining attendance to follow-up care? The Swiss childhood cancer survivor study. Psychooncology. 2011 Oct;20(10):1034-43. doi: 10.1002/pon.1823. Epub 2010 Aug 4. PMID 20687196
- [Result] Michel G, Rebholz CE, von der Weid NX, Bergstraesser E, Kuehni CE. Psychological distress in adult survivors of childhood cancer: the Swiss Childhood Cancer Survivor study. J Clin Oncol. 2010 Apr 1;28(10):1740-8. doi: 10.1200/JCO.2009.23.4534. Epub 2010 Mar 1. PMID 20194864
- [Result] Michel G, Gianinazzi ME, Eiser C, Bergstraesser E, Vetsch J, von der Weid N, Kuehni CE; Swiss Paediatric Oncology Group. Preferences for long-term follow-up care in childhood cancer survivors. Eur J Cancer Care (Engl). 2016 Nov;25(6):1024-1033. doi: 10.1111/ecc.12560. Epub 2016 Aug 23. PMID 27550385
- [Result] Rebholz CE, Rueegg CS, Michel G, Ammann RA, von der Weid NX, Kuehni CE, Spycher BD; Swiss Paediatric Oncology Group (SPOG). Clustering of health behaviours in adult survivors of childhood cancer and the general population. Br J Cancer. 2012 Jul 10;107(2):234-42. doi: 10.1038/bjc.2012.250. Epub 2012 Jun 21. PMID 22722311
- [Result] Marquis A, Strippoli MP, Spycher BD, Rebholz CE, von der Weid NX, Kuehni CE; Swiss Pediatric Oncology Group. Paracetamol, nonsteroidal anti-inflammatory drugs, and risk of asthma in adult survivors of childhood cancer. J Allergy Clin Immunol. 2011 Jan;127(1):270-2. doi: 10.1016/j.jaci.2010.08.044. Epub 2010 Nov 18. No abstract available. PMID 21093027
- [Result] Belle FN, Kasteler R, Schindera C, Bochud M, Ammann RA, von der Weid NX, Kuehni CE; Swiss Pediatric Oncology Group (SPOG). No evidence of overweight in long-term survivors of childhood cancer after glucocorticoid treatment. Cancer. 2018 Sep 1;124(17):3576-3585. doi: 10.1002/cncr.31599. Epub 2018 Aug 17. PMID 30119140
- [Result] Belle FN, Wenke-Zobler J, Cignacco E, Spycher BD, Ammann RA, Kuehni CE, Zimmermann K. Overweight in childhood cancer patients at diagnosis and throughout therapy: A multicentre cohort study. Clin Nutr. 2019 Apr;38(2):835-841. doi: 10.1016/j.clnu.2018.02.022. Epub 2018 Mar 2. PMID 29544999
- [Result] Belle FN, Weiss A, Schindler M, Goutaki M, Bochud M, Zimmermann K, von der Weid N, Ammann RA, Kuehni CE. Overweight in childhood cancer survivors: the Swiss Childhood Cancer Survivor Study. Am J Clin Nutr. 2018 Jan 1;107(1):3-11. doi: 10.1093/ajcn/nqx006. PMID 29381792
- [Result] Kasteler R, Belle F, Schindera C, Barben J, Gumy-Pause F, Tinner EM, Kuehni CE; Swiss Pediatric Oncology Group (SPOG). Prevalence and reasons for smoking in adolescent Swiss childhood cancer survivors. Pediatr Blood Cancer. 2019 Jan;66(1):e27438. doi: 10.1002/pbc.27438. Epub 2018 Sep 21. PMID 30239111
- [Result] Clemens E, van den Heuvel-Eibrink MM, Mulder RL, Kremer LCM, Hudson MM, Skinner R, Constine LS, Bass JK, Kuehni CE, Langer T, van Dalen EC, Bardi E, Bonne NX, Brock PR, Brooks B, Carleton B, Caron E, Chang KW, Johnston K, Knight K, Nathan PC, Orgel E, Prasad PK, Rottenberg J, Scheinemann K, de Vries ACH, Walwyn T, Weiss A, Am Zehnhoff-Dinnesen A, Cohn RJ, Landier W; International Guideline Harmonization Group ototoxicity group. Recommendations for ototoxicity surveillance for childhood, adolescent, and young adult cancer survivors: a report from the International Late Effects of Childhood Cancer Guideline Harmonization Group in collaboration with the PanCare Consortium. Lancet Oncol. 2019 Jan;20(1):e29-e41. doi: 10.1016/S1470-2045(18)30858-1. PMID 30614474
- [Result] Reulen RC, Wong KF, Bright CJ, Winter DL, Alessi D, Allodji RM, Bagnasco F, Bardi E, Bautz A, Byrne J, Feijen EA, Fidler-Benaoudia MM, Diallo I, Garwicz S, Grabow D, Gudmundsdottir T, Guha J, Haddy N, Hogsholt S, Jankovic M, Kaatsch P, Kaiser M, Kuonen R, Linge H, Ofstaas H, Ronckers CM, Hau EM, Skinner R, van Leeuwen FE, Teepen JC, Veres C, Zrafi W, Debiche G, Llanas D, Terenziani M, Vu-Bezin G, Wesenberg F, Wiebe T, Sacerdote C, Jakab Z, Haupt R, Lahteenmaki PM, Zadravec Zaletel L, Kuehni CE, Winther JF, de Vathaire F, Kremer LC, Hjorth L, Hawkins MM. Risk of digestive cancers in a cohort of 69 460 five-year survivors of childhood cancer in Europe: the PanCareSurFup study. Gut. 2020 Nov 2:gutjnl-2020-322237. doi: 10.1136/gutjnl-2020-322237. Online ahead of print. PMID 33139271
- [Result] Otth M, Schindera C, Gungor T, Ansari M, Scheinemann K, Belle FN, Latzin P, von der Weid N, Kuehni CE; Swiss Pediatric Oncology Group (SPOG). Transplant characteristics and self-reported pulmonary outcomes in Swiss childhood cancer survivors after hematopoietic stem cell transplantation-a cohort study. Bone Marrow Transplant. 2021 May;56(5):1065-1076. doi: 10.1038/s41409-020-01137-1. Epub 2020 Nov 25. PMID 33239655
- [Result] Norsker FN, Pedersen C, Armstrong GT, Robison LL, McBride ML, Hawkins M, Kuehni CE, de Vathaire F, Berbis J, Kremer LC, Haupt R, Kenborg L, Winther JF. Late Effects in Childhood Cancer Survivors: Early Studies, Survivor Cohorts, and Significant Contributions to the Field of Late Effects. Pediatr Clin North Am. 2020 Dec;67(6):1033-1049. doi: 10.1016/j.pcl.2020.07.002. PMID 33131533
- [Result] Langer T, Clemens E, Broer L, Maier L, Uitterlinden AG, de Vries ACH, van Grotel M, Pluijm SFM, Binder H, Mayer B, von dem Knesebeck A, Byrne J, van Dulmen-den Broeder E, Crocco M, Grabow D, Kaatsch P, Kaiser M, Spix C, Kenborg L, Winther JF, Rechnitzer C, Hasle H, Kepak T, van der Kooi AF, Kremer LC, Kruseova J, Bielack S, Sorg B, Hecker-Nolting S, Kuehni CE, Ansari M, Kompis M, van der Pal H, Parfitt R, Deuster D, Matulat P, Tillmanns A, Tissing WJE, Beck JD, Elsner S, Am Zehnhoff-Dinnesen A, van den Heuvel-Eibrink MM, Zolk O; PanCareLIFE consortium. Usefulness of current candidate genetic markers to identify childhood cancer patients at risk for platinum-induced ototoxicity: Results of the European PanCareLIFE cohort study. Eur J Cancer. 2020 Oct;138:212-224. doi: 10.1016/j.ejca.2020.07.019. Epub 2020 Sep 6. PMID 32905960
- [Result] Winther JF, Kenborg L, Byrne J, Hjorth L, Kaatsch P, Kremer LC, Kuehni CE, Auquier P, Michel G, de Vathaire F, Haupt R, Skinner R, Madanat-Harjuoja LM, Tryggvadottir L, Wesenberg F, Reulen RC, Grabow D, Ronckers CM, van Dulmen-den Broeder E, van den Heuvel-Eibrink MM, Schindler M, Berbis J, Holmqvist AS, Gudmundsdottir T, de Fine Licht S, Bonnesen TG, Asdahl PH, Bautz A, Kristoffersen AK, Himmerslev L, Hasle H, Olsen JH, Hawkins MM. Childhood cancer survivor cohorts in Europe. Acta Oncol. 2015 May;54(5):655-68. doi: 10.3109/0284186X.2015.1008648. Epub 2015 Mar 27. PMID 25813473
- [Result] Bhatia S, Armenian SH, Armstrong GT, van Dulmen-den Broeder E, Hawkins MM, Kremer LC, Kuehni CE, Olsen JH, Robison LL, Hudson MM. Collaborative Research in Childhood Cancer Survivorship: The Current Landscape. J Clin Oncol. 2015 Sep 20;33(27):3055-64. doi: 10.1200/JCO.2014.59.8052. Epub 2015 Aug 24. PMID 26304891
- [Result] Hjorth L, Haupt R, Skinner R, Grabow D, Byrne J, Karner S, Levitt G, Michel G, van der Pal H, Bardi E, Beck JD, de Vathaire F, Essig S, Frey E, Garwicz S, Hawkins M, Jakab Z, Jankovic M, Kazanowska B, Kepak T, Kremer L, Lackner H, Sugden E, Terenziani M, Zaletel LZ, Kaatsch P; PanCare Network. Survivorship after childhood cancer: PanCare: a European Network to promote optimal long-term care. Eur J Cancer. 2015 Jul;51(10):1203-11. doi: 10.1016/j.ejca.2015.04.002. Epub 2015 May 6. PMID 25958037
- [Result] Brown MC, Levitt GA, Frey E, Bardi E, Haupt R, Hjorth L, Kremer L, Kuehni CE, Lettner C, Mulder RL, Michel G, Skinner R; PanCareSurFup Consortium. The views of European clinicians on guidelines for long-term follow-up of childhood cancer survivors. Pediatr Blood Cancer. 2015 Feb;62(2):322-328. doi: 10.1002/pbc.25310. Epub 2014 Nov 8. PMID 25382221
- [Result] Feijen EA, Font-Gonzalez A, van Dalen EC, van der Pal HJ, Reulen RC, Winter DL, Kuehni CE, Haupt R, Alessi D, Byrne J, Bardi E, Jakab Z, Grabow D, Garwicz S, Jankovic M, Levitt GA, Skinner R, Zadravec Zaletel L, Hjorth L, Tissing WJ, de Vathaire F, Hawkins MM, Kremer LC; PanCareSurFup consortium. Late Cardiac Events after Childhood Cancer: Methodological Aspects of the Pan-European Study PanCareSurFup. PLoS One. 2016 Sep 19;11(9):e0162778. doi: 10.1371/journal.pone.0162778. eCollection 2016. PMID 27643694
- [Result] Adam M, Rueegg CS, Schmidlin K, Spoerri A, Niggli F, Grotzer M, von der Weid NX, Egger M, Probst-Hensch N, Zwahlen M, Kuehni CE; Swiss Paediatric Oncology Group; Swiss National Cohort Study. Socioeconomic disparities in childhood cancer survival in Switzerland. Int J Cancer. 2016 Jun 15;138(12):2856-66. doi: 10.1002/ijc.30029. Epub 2016 Mar 1. PMID 26840758
- [Result] Byrne J, Alessi D, Allodji RS, Bagnasco F, Bardi E, Bautz A, Bright CJ, Brown M, Diallo I, Feijen EAML, Fidler MM, Frey E, Garwicz S, Grabow D, Gudmundsdottir T, Hagberg O, Harila-Saari A, Hau EM, Haupt R, Hawkins MM, Jakab Z, Jankovic M, Kaatsch P, Kaiser M, Kremer LCM, Kuehni CE, Kuonen R, Ladenstein R, Lahteenmaki PM, Levitt G, Linge H, LLanas D, Michel G, Morsellino V, Mulder RL, Reulen RC, Ronckers CM, Sacerdote C, Skinner R, Steliarova-Foucher E, van der Pal HJ, de Vathaire F, Vu Bezin G, Wesenberg F, Wiebe T, Winter DL, Winther JF, Witthoff E, Zadravec Zaletel L, Hjorth L. The PanCareSurFup consortium: research and guidelines to improve lives for survivors of childhood cancer. Eur J Cancer. 2018 Nov;103:238-248. doi: 10.1016/j.ejca.2018.08.017. Epub 2018 Oct 1. PMID 30286417
- [Result] Byrne J, Grabow D, Campbell H, O'Brien K, Bielack S, Am Zehnhoff-Dinnesen A, Calaminus G, Kremer L, Langer T, van den Heuvel-Eibrink MM, van Dulmen-den Broeder E, Baust K, Bautz A, Beck JD, Berger C, Binder H, Borgmann-Staudt A, Broer L, Cario H, Casagranda L, Clemens E, Deuster D, de Vries A, Dirksen U, Winther JF, Fossa S, Font-Gonzalez A, Grandage V, Haupt R, Hecker-Nolting S, Hjorth L, Kaiser M, Kenborg L, Kepak T, Kepakova K, Knudsen LE, Krawczuk-Rybak M, Kruseova J, Kuehni CE, Kunstreich M, Kuonen R, Lackner H, Leiper A, Loeffen EAH, Luks A, Modan-Moses D, Mulder R, Parfitt R, Paul NW, Ranft A, Ruud E, Schilling R, Spix C, Stefanowicz J, Straubeta G, Uitterlinden AG, van den Berg M, van der Kooi AL, van Dijk M, van Leeuwen F, Zolk O, Zoller D, Kaatsch P; PanCareLIFE consortium. PanCareLIFE: The scientific basis for a European project to improve long-term care regarding fertility, ototoxicity and health-related quality of life after cancer occurring among children and adolescents. Eur J Cancer. 2018 Nov;103:227-237. doi: 10.1016/j.ejca.2018.08.007. Epub 2018 Sep 29. PMID 30273888
- [Result] Fidler MM, Reulen RC, Winter DL, Allodji RS, Bagnasco F, Bardi E, Bautz A, Bright CJ, Byrne J, Feijen EAM, Garwicz S, Grabow D, Gudmundsdottir T, Guha J, Haddy N, Jankovic M, Kaatsch P, Kaiser M, Kuonen R, Linge H, Maule M, Merletti F, Ofstaas H, Ronckers CM, Skinner R, Teepen J, Terenziani M, Vu-Bezin G, Wesenberg F, Wiebe T, Jakab Z, Haupt R, Lahteenmaki P, Zaletel LZ, Kuehni CE, Winther JF, de Vathaire F, Kremer LC, Hjorth L, Hawkins MM. Risk of Subsequent Bone Cancers Among 69 460 Five-Year Survivors of Childhood and Adolescent Cancer in Europe. J Natl Cancer Inst. 2018 Feb 1;110(2). doi: 10.1093/jnci/djx165. PMID 28954302
- [Result] Grabow D, Kaiser M, Hjorth L, Byrne J, Alessi D, Allodji RS, Bagnasco F, Bardi E, Bautz A, Bright CJ, de Vathaire F, Feijen EAM, Garwicz S, Hagberg O, Haupt R, Hawkins MM, Jakab Z, Kremer LCM, Kuehni CE, Kuonen R, Lahteenmaki PM, Reulen RC, Ronckers CM, Sacerdote C, Vu-Bezin G, Wesenberg F, Wiebe T, Winter DL, Winther JF, Zaletel LZ, Kaatsch P; PanCareSurFup Consortium. The PanCareSurFup cohort of 83,333 five-year survivors of childhood cancer: a cohort from 12 European countries. Eur J Epidemiol. 2018 Mar;33(3):335-349. doi: 10.1007/s10654-018-0370-3. Epub 2018 Mar 2. PMID 29497894
- [Result] Weiss A, Kuonen R, Brockmeier H, Grotzer M, Candreia C, Maire R, Senn P, Stieger C, Rosenfeld J, Veraguth D, Kompis M, Scheinemann K, Kuehni CE; Swiss Pediatric Oncology Group (SPOG). Audiological monitoring in Swiss childhood cancer patients. Pediatr Blood Cancer. 2018 Mar;65(3). doi: 10.1002/pbc.26877. Epub 2017 Dec 12. PMID 29230928
- [Result] Jankovic M, Haupt R, Spinetta JJ, Beck JD, Byrne J, Calaminus G, Lackner H, Biondi A, Oeffinger K, Hudson M, Skinner R, Reaman G, van der Pal H, Kremer L, den Hartogh J, Michel G, Frey E, Bardi E, Hawkins M, Rizvi K, Terenziani M, Valsecchi MG, Bode G, Jenney M, de Vathaire F, Garwicz S, Levitt GA, Grabow D, Kuehni CE, Schrappe M, Hjorth L; participants in PanCare. Long-term survivors of childhood cancer: cure and care-the Erice Statement (2006) revised after 10 years (2016). J Cancer Surviv. 2018 Oct;12(5):647-650. doi: 10.1007/s11764-018-0701-0. Epub 2018 Jun 26. PMID 29946794
- [Result] Bright CJ, Hawkins MM, Winter DL, Alessi D, Allodji RS, Bagnasco F, Bardi E, Bautz A, Byrne J, Feijen EAM, Fidler MM, Garwicz S, Grabow D, Gudmundsdottir T, Guha J, Haddy N, Jankovic M, Kaatsch P, Kaiser M, Kuehni CE, Linge H, Ofstaas H, Ronckers CM, Skinner R, Teepen JC, Terenziani M, Vu-Bezin G, Wesenberg F, Wiebe T, Sacerdote C, Jakab Z, Haupt R, Lahteenmaki P, Zaletel LZ, Kuonen R, Winther JF, de Vathaire F, Kremer LC, Hjorth L, Reulen RC; PanCareSurFup Consortium. Risk of Soft-Tissue Sarcoma Among 69 460 Five-Year Survivors of Childhood Cancer in Europe. J Natl Cancer Inst. 2018 Jun 1;110(6):649-660. doi: 10.1093/jnci/djx235. PMID 29165710
- [Result] Kasteler R, Kam LMH, Weiss A, Waespe N, Sommer G, Singer F, von der Weid NX, Ansari M, Kuehni CE; Swiss Pediatric Oncology Group (SPOG). Monitoring pulmonary health in Swiss childhood cancer survivors. Pediatr Blood Cancer. 2018 Oct;65(10):e27255. doi: 10.1002/pbc.27255. Epub 2018 Jun 15. PMID 29905401
- [Result] Tonorezos ES, Barnea D, Cohn RJ, Cypriano MS, Fresneau BC, Haupt R, Hjorth L, Ishida Y, Kruseova J, Kuehni CE, Kurkure PA, Langer T, Nathan PC, Skeen JE, Skinner R, Tacyildiz N, van den Heuvel-Eibrink MM, Winther JF, Hudson MM, Oeffinger KC. Models of Care for Survivors of Childhood Cancer From Across the Globe: Advancing Survivorship Care in the Next Decade. J Clin Oncol. 2018 Jul 20;36(21):2223-2230. doi: 10.1200/JCO.2017.76.5180. Epub 2018 Jun 6. PMID 29874138
- [Result] Allodji RS, Hawkins MM, Bright CJ, Fidler-Benaoudia MM, Winter DL, Alessi D, Fresneau B, Journy N, Morsellino V, Bardi E, Bautz A, Byrne J, Feijen ELA, Teepen JC, Vu-Bezin G, Rubino C, Garwicz S, Grabow D, Gudmundsdottir T, Guha J, Hau EM, Jankovic M, Kaatsch P, Kaiser M, Linge H, Muraca M, Llanas D, Veres C, Ofstaas H, Diallo I, Mansouri I, Ronckers CM, Skinner R, Terenziani M, Wesenberg F, Wiebe T, Sacerdote C, Jakab Z, Haupt R, Lahteenmaki P, Zaletel LZ, Kuehni CE, Winther JF, Michel G, Kremer LCM, Hjorth L, Haddy N, de Vathaire F, Reulen RC. Risk of subsequent primary leukaemias among 69,460 five-year survivors of childhood cancer diagnosed from 1940 to 2008 in Europe: A cohort study within PanCareSurFup. Eur J Cancer. 2019 Aug;117:71-83. doi: 10.1016/j.ejca.2019.05.013. Epub 2019 Jun 28. PMID 31260818
- [Result] Weiss A, Sommer G, Schindera C, Wengenroth L, Karow A, Diezi M, Michel G, Kuehni CE; Swiss Paediatric Oncology Group (SPOG). Hearing loss and quality of life in survivors of paediatric CNS tumours and other cancers. Qual Life Res. 2019 Feb;28(2):515-521. doi: 10.1007/s11136-018-2021-2. Epub 2018 Oct 10. PMID 30306534
- [Result] Essig S, Michel G, Dupont C, Kiss A, Bergstraesser E, Tinner EM, Kuehni CE; Swiss Pediatric Oncology Group (SPOG). Communicating "cure" to pediatric oncology patients: A mixed-methods study. Pediatr Blood Cancer. 2019 Jun;66(6):e27661. doi: 10.1002/pbc.27661. Epub 2019 Feb 7. PMID 30729685
- [Result] Hau EM, Caccia JN, Kasteler R, Spycher B, Suter T, Ammann RA, von der Weid NX, Kuehni CE. Cardiovascular disease after childhood acute lymphoblastic leukaemia: a cohort study. Swiss Med Wkly. 2019 Mar 10;149:w20012. doi: 10.4414/smw.2019.20012. eCollection 2019 Feb 25. PMID 30852834
- [Result] Belle FN, Beck Popovic M, Ansari M, Otth M, Kuehni CE, Bochud M. Nutritional Assessment of Childhood Cancer Survivors (the Swiss Childhood Cancer Survivor Study-Nutrition): Protocol for a Multicenter Observational Study. JMIR Res Protoc. 2019 Nov 18;8(11):e14427. doi: 10.2196/14427. PMID 31738177
- [Result] Belle FN, Schindera C, Guessous I, Popovic MB, Ansari M, Kuehni CE, Bochud M. Sodium and Potassium Intakes and Cardiovascular Risk Profiles in Childhood Cancer Survivors: The SCCSS-Nutrition Study. Nutrients. 2019 Dec 24;12(1):57. doi: 10.3390/nu12010057. PMID 31878342
- [Result] Schindera C, Weiss A, Hagenbuch N, Otth M, Diesch T, von der Weid N, Kuehni CE; Swiss Pediatric Oncology Group (SPOG). Physical activity and screen time in children who survived cancer: A report from the Swiss Childhood Cancer Survivor Study. Pediatr Blood Cancer. 2020 Feb;67(2):e28046. doi: 10.1002/pbc.28046. Epub 2019 Nov 20. PMID 31750617
- [Result] Langer T, Clemens E, Broer L, Maier L, Uitterlinden AG, de Vries ACH, van Grotel M, Pluijm SFM, Binder H, Mayer B, von dem Knesebeck A, Byrne J, van Dulmen-den Broeder E, Crocco M, Grabow D, Kaatsch P, Kaiser M, Spix C, Kenborg L, Winther JF, Rechnitzer C, Hasle H, Kepak T, van der Kooi AF, Kremer LC, Kruseova J, Bielack S, Sorg B, Hecker-Nolting S, Kuehni CE, Ansari M, Kompis M, van der Pal HJ, Parfitt R, Deuster D, Matulat P, Tillmanns A, Tissing WJE, Beck JD, Elsner S, Am Zehnhoff-Dinnesen A, van den Heuvel-Eibrink MM, Zolk O; PanCareLIFE consortium. Association of candidate pharmacogenetic markers with platinum-induced ototoxicity: PanCareLIFE dataset. Data Brief. 2020 Aug 24;32:106227. doi: 10.1016/j.dib.2020.106227. eCollection 2020 Oct. PMID 32939381
- [Result] Waespe N, Belle FN, Redmond S, Schindera C, Spycher BD, Rossler J, Ansari M, Kuehni CE; Swiss Paediatric Oncology Group (SPOG). Cancer predisposition syndromes as a risk factor for early second primary neoplasms after childhood cancer - A national cohort study. Eur J Cancer. 2021 Mar;145:71-80. doi: 10.1016/j.ejca.2020.11.042. Epub 2021 Jan 7. PMID 33423008
- [Result] Waespe N, Strebel S, Marino D, Mattiello V, Muet F, Nava T, Schindera C, Belle FN, Mader L, Spoerri A, Kuehni CE, Ansari M. Predictors for participation in DNA self-sampling of childhood cancer survivors in Switzerland. BMC Med Res Methodol. 2021 Oct 30;21(1):236. doi: 10.1186/s12874-021-01428-1. PMID 34717553
- [Result] Belle FN, Chatelan A, Kasteler R, Mader L, Guessous I, Beck-Popovic M, Ansari M, Kuehni CE, Bochud M. Dietary Intake and Diet Quality of Adult Survivors of Childhood Cancer and the General Population: Results from the SCCSS-Nutrition Study. Nutrients. 2021 May 22;13(6):1767. doi: 10.3390/nu13061767. PMID 34067298
- [Result] Dudley IM, Sunguc C, Heymer EJ, Winter DL, Teepen JC, Belle FN, Bardi E, Bagnasco F, Gudmundsdottir T, Skinner R, Michel G, Byrne J, Ofstaas H, Jankovic M, Mazic MC, Mader L, Loonen J, Garwicz S, Wiebe T, Alessi D, Allodji RS, Haddy N, Grabow D, Kaatsch P, Kaiser M, Maule MM, Jakab Z, Gunnes MW, Terenziani M, Zaletel LZ, Kuehni CE, Haupt R, de Vathaire F, Kremer LC, Lahteenmaki PM, Winther JF, Hjorth L, Hawkins MM, Reulen RC. Risk of subsequent primary lymphoma in a cohort of 69,460 five-year survivors of childhood and adolescent cancer in Europe: The PanCareSurFup study. Cancer. 2023 Feb 1;129(3):426-440. doi: 10.1002/cncr.34561. Epub 2022 Nov 29. PMID 36444554
- [Result] Sunguc C, Hawkins MM, Winter DL, Dudley IM, Heymer EJ, Teepen JC, Allodji RS, Belle FN, Bagnasco F, Byrne J, Bardi E, Ronckers CM, Haddy N, Gudmundsdottir T, Garwicz S, Jankovic M, van der Pal HJH, Mazic MC, Schindera C, Grabow D, Maule MM, Kaatsch P, Kaiser M, Fresneau B, Michel G, Skinner R, Wiebe T, Sacerdote C, Jakab Z, Gunnes MW, Terenziani M, Winther JF, Lahteenmaki PM, Zaletel LZ, Kuehni CE, Kremer LC, Haupt R, de Vathaire F, Hjorth L, Reulen RC. Risk of subsequent primary oral cancer in a cohort of 69,460 5-year survivors of childhood and adolescent cancer in Europe: the PanCareSurFup study. Br J Cancer. 2023 Jan;128(1):80-90. doi: 10.1038/s41416-022-02016-w. Epub 2022 Nov 1. PMID 36319851
- [Result] Otth M, Yammine S, Usemann J, Latzin P, Mader L, Spycher B, Gungor T, Scheinemann K, Kuehni CE; Swiss Pediatric Oncology Group (SPOG). Longitudinal lung function in childhood cancer survivors after hematopoietic stem cell transplantation. Bone Marrow Transplant. 2022 Feb;57(2):207-214. doi: 10.1038/s41409-021-01509-1. Epub 2021 Nov 8. PMID 34750563
- [Result] Strebel S, Mader L, Slama T, Waespe N, Weiss A, Parfitt R, Am Zehnhoff-Dinnesen A, Kompis M, von der Weid NX, Ansari M, Kuehni CE. Severity of hearing loss after platinum chemotherapy in childhood cancer survivors. Pediatr Blood Cancer. 2022 Sep;69(9):e29755. doi: 10.1002/pbc.29755. Epub 2022 Jun 19. PMID 35723448
- [Result] Mader L, Slama T, Schindera C, Rossler J, von der Weid NX, Belle FN, Kuehni CE. Social, emotional, and behavioral functioning in young childhood cancer survivors with chronic health conditions. Pediatr Blood Cancer. 2022 Sep;69(9):e29756. doi: 10.1002/pbc.29756. Epub 2022 May 13. PMID 35561093
- [Result] Belle FN, Schindera C, Ansari M, Armstrong GT, Beck-Popovic M, Howell R, Leisenring WM, Meacham LR, Rossler J, Spycher BD, Tonorezos E, von der Weid NX, Yasui Y, Oeffinger KC, Kuehni CE. Risk factors for overweight and obesity after childhood acute lymphoblastic leukemia in North America and Switzerland: A comparison of two cohort studies. Cancer Med. 2023 Oct;12(20):20423-20436. doi: 10.1002/cam4.6588. Epub 2023 Oct 9. PMID 37807946
- [Result] Wang Y, Ronckers CM, van Leeuwen FE, Moskowitz CS, Leisenring W, Armstrong GT, de Vathaire F, Hudson MM, Kuehni CE, Arnold MA, Demoor-Goldschmidt C, Green DM, Henderson TO, Howell RM, Ehrhardt MJ, Neglia JP, Oeffinger KC, van der Pal HJH, Robison LL, Schaapveld M, Turcotte LM, Waespe N, Kremer LCM, Teepen JC; International Consortium for Pooled Studies on Subsequent Malignancies after Childhood and Adolescent Cancer. Subsequent female breast cancer risk associated with anthracycline chemotherapy for childhood cancer. Nat Med. 2023 Sep;29(9):2268-2277. doi: 10.1038/s41591-023-02514-1. Epub 2023 Sep 11. PMID 37696934
- [Result] Baenziger J, Roser K, Mader L, Ilic A, Sansom-Daly UM, von Bueren AO, Tinner EM, Michel G. Post-traumatic growth in parents of long-term childhood cancer survivors compared to the general population: A report from the Swiss childhood cancer survivor study-Parents. Psychooncology. 2024 Jan;33(1):e6246. doi: 10.1002/pon.6246. Epub 2023 Dec 4. PMID 38047716
- [Result] Christen S, Roser K, Mader L, Otth M, Scheinemann K, Sommer G, Kuehni C, Michel G. Incidence and prevalence of musculoskeletal health conditions in survivors of childhood and adolescent cancers: A report from the Swiss childhood cancer survivor study. Cancer Med. 2024 Apr;13(8):e7204. doi: 10.1002/cam4.7204. PMID 38650581
- [Result] Hau EM, Slama T, Essig S, Michel G, Wengenroth L, Bergstraesser E, von der Weid NX, Schindera C, Kuehni CE. Validation of self-reported cardiovascular problems in childhood cancer survivors by contacting general practitioners: feasibility and results. BMC Prim Care. 2024 Mar 8;25(1):81. doi: 10.1186/s12875-024-02322-7. PMID 38459512
- [Result] Raguindin PF, Rueegg CS, Kalin S, Bergstraesser E, von der Weid NX, Tinner EM, Kuehni CE, Michel G. Longitudinal changes of psychological distress among childhood cancer survivors: The Swiss Childhood Cancer Survivor Study. Pediatr Blood Cancer. 2024 Aug;71(8):e31095. doi: 10.1002/pbc.31095. Epub 2024 Jun 2. PMID 38825751
- [Result] Slama T, Mader L, Zarkovic M, Malar R, Schifferli A, von der Weid NX, Kuehni CE, Schindera C. Chronic health conditions after childhood Langerhans cell histiocytosis: Results from the Swiss Childhood Cancer Survivor Study. J Cancer Surviv. 2025 Aug;19(4):1212-1221. doi: 10.1007/s11764-024-01544-z. Epub 2024 Feb 14. PMID 38353855
- [Result] Zarkovic M, Sommer G, Nigg C, Slama T, Schneider C, Ansari M, von der Weid N, Schindera C, Kuehni CE. Parental smoking and respiratory outcomes in young childhood cancer survivors. Pediatr Blood Cancer. 2024 Nov;71(11):e31310. doi: 10.1002/pbc.31310. Epub 2024 Sep 3. PMID 39228077
- [Result] Nigg C, Matti C, Jorger P, von Bueren AO, Filippi C, Diesch-Furlanetto T, Tomasikova Z, Kuehni CE, Sommer G. Dental Health of Childhood Cancer Survivors-A Report From the Swiss Childhood Cancer Survivor Study (SCCSS). Pediatr Blood Cancer. 2025 May;72(5):e31629. doi: 10.1002/pbc.31629. Epub 2025 Mar 6. PMID 40051213
- See also: Swiss Childhood Cancer Registry — https://childhoodcancerregistry.ch
- See also: Swiss Childhood Cancer Survivor Study, SCCSS — https://www.swiss-ccss.ch